CLINICAL TRIAL: NCT03797924
Title: Intercostobrachial Nerve Block (ICBN) for Tourniquet Pain: Is it Necessary?
Acronym: ICBN
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB201802525; OCR19802 (Other: OnCore)
Record Dates: First submitted 2019-01-01; First posted 2019-01-09 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Nerve Block; Pain
Keywords: Intercostobrachial Nerve Block; Tourniquet Pain; Upper Limb Surgeries
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive ICBN with ropivacaine or no ICBN or ropivacaine.
Who Masked: Participant, Care Provider
Masking Description: In order to blind anesthesia providers in the room and nurses in Post-op Anesthesia Care Unit (PACU), the site of injection for ICBN will be prepped with tinted chlorhexidine in all patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICBN with ropivacaine (Active Comparator): Participants will receive ICBN with ropivacaine. In order to blind anesthesia providers in the room and nurses in PACU, the site of injection for ICBN will be prepped with tinted chlorhexidine in all patients.
  Interventions: Drug: Receive ICBN with ropivacaine
- No ICBN block (Placebo Comparator): Participants will have the site prepped, but no ICBN block given. In order to blind anesthesia providers in the room and nurses in PACU, the site of injection for ICBN will be prepped with tinted chlorhexidine in all patients.
  Interventions: Behavioral: No ICBN block

INTERVENTIONS:
Drug: Receive ICBN with ropivacaine — ICBN block will be performed using US guidance depositing 10 ml of 0.5% ropivacaine in the plane between pectoralis minor and serratus anterior over the 2nd and 3rd intercostal space.
  Other Names: Naropin
  Arms: ICBN with ropivacaine
Behavioral: No ICBN block — The site of injection will be prepped with tinted chlorhexidine
  Arms: No ICBN block

SUMMARY:
In this study the investigators would like to show that when patients undergo upper limb surgery under supraclavicular brachial plexus block, additional blocking of the Intercostobrachial Nerve Block (ICBN) does not affect the incidence or course of tourniquet pain.

DETAILED DESCRIPTION:
The ICBN is a cutaneous sensory nerve that supplies the medial aspect of the upper arm. Traditionally this nerve is blocked to alleviate tourniquet pain. The etiology of tourniquet pain is complex and the study team hypothesize that blocking the ICBN has no impact on tourniquet pain. Patients will receive a supraclavicular block and be divided into two groups; ICBN with local anesthetic or ICBN with saline. All patients in this study will receive a supraclavicular block as their primary anesthetic and then be divided into two groups; those who receive ICBN and those who do not. Amount of intraoperative analgesics, conversion to deep sedation or general anesthesia, and onset of time to tourniquet pain will be the primary measures of this study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) 1-3
* Distal upper extremity surgery with anticipated use of tourniquet
* Outpatient surgery
* Patients who desire regional anesthesia as primary anesthetic

Exclusion Criteria:

* ASA 4 or greater
* Allergies to local anesthetic
* Refusal of regional anesthesia
* History of chronic pain syndromes
* Patients who do not desire regional anesthesia as primary anesthetic

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Change between the 2 groups assessed by the incidence of tourniquet pain reported by the patient on a Descriptor Differential Scale of Pain Intensity (DDSI) | From intraoperative pre tourniquet insufflation to intraoperative release of tourniquet (up to 2 hours)
  Tourniquet pain defined by the presence of dull or aching pain underneath the tourniquet

SECONDARY OUTCOMES:
Change between the 2 groups depth of anesthesia during surgery to alleviate tourniquet pain as assessed by the American Society of Anesthesiologist (ASA) Continuum of Depth of Sedation definition of general anesthesia and levels of sedation/analgesia. | From intraoperative pre tourniquet insufflation to intraoperative release of tourniquet (up to 2 hours)
  Determine required depth of anesthesia during surgery to alleviate tourniquet pain
Change between the 2 groups assessed by intraoperative opioid consumption | From intraoperative pre tourniquet insufflation to intraoperative release of tourniquet (up to 2 hours)
  Determine amount of intraoperative opioid consumption due to tourniquet pain
Change between the 2 groups assessed by time to onset of tourniquet pain | From intraoperative pre tourniquet insufflation to intraoperative release of tourniquet (up to 2 hours)
  Determine the time to onset of tourniquet pain
Change between the 2 groups in reported severity of tourniquet pain | From intraoperative pre tourniquet insufflation to intraoperative release of tourniquet (up to 2 hours)
  Determine if ICBN has an affect on the severity of tourniquet pain as assessed by Descriptor Differential Scale of Pain Intensity (DDSI) There are 10 points along which patients can rate their pain intensity to the right and left of each descriptor, so the pain is rated on a 21 point scale for each descriptor. Pain intensity is defined as a mean of the ratings and can range from 0 to 20.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Le-Wendling, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Satsumae T, Yamaguchi H, Inomata S, Tanaka M. Magnesium sulfate attenuates tourniquet pain in healthy volunteers. J Anesth. 2013 Apr;27(2):231-5. doi: 10.1007/s00540-012-1493-4. Epub 2012 Oct 7. PMID 23053464
- [Result] Hagenouw RR, Bridenbaugh PO, van Egmond J, Stuebing R. Tourniquet pain: a volunteer study. Anesth Analg. 1986 Nov;65(11):1175-80. PMID 3767015
- [Result] Valli H, Rosenberg PH, Kytta J, Nurminen M. Arterial hypertension associated with the use of a tourniquet with either general or regional anaesthesia. Acta Anaesthesiol Scand. 1987 May;31(4):279-83. doi: 10.1111/j.1399-6576.1987.tb02566.x. PMID 3591250
- [Result] Crews JC, Cahall M, Behbehani MM. The neurophysiologic mechanisms of tourniquet pain. The activity of neurons in the rostroventral medulla in the rat. Anesthesiology. 1994 Sep;81(3):730-6. doi: 10.1097/00000542-199409000-00027. PMID 8092519
- [Result] MacIver MB, Tanelian DL. Activation of C fibers by metabolic perturbations associated with tourniquet ischemia. Anesthesiology. 1992 Apr;76(4):617-23. doi: 10.1097/00000542-199204000-00020. PMID 1550287
- [Result] Tschaikowsky K, Hemmerling T. Comparison of the effect of EMLA and semicircular subcutaneous anaesthesia in the prevention of tourniquet pain during plexus block anaesthesia of the arm. Anaesthesia. 1998 Apr;53(4):390-3. doi: 10.1046/j.1365-2044.1998.00301.x. PMID 9613307